CLINICAL TRIAL: NCT05614349
Title: Canadian Adaptive Platform Trial of Treatments for COVID-19 in Community Settings
Acronym: CanTreatCOVID
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Health Canada (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTO 4133
Record Dates: First submitted 2022-11-09; First posted 2022-11-14 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination; Antioxidants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Paxlovid (Experimental): Nirmatrelvir/ritonavir (Paxlovid™) BD x 5 days (this arm has been closed of Sept 30th 2024)
  Interventions: Drug: Paxlovid
- Control group (No Intervention): Usual care (i.e., supportive care and symptom relief)
- Antioxidant Therapy - Intervention (arm 3) (Experimental): Antioxidant therapy (comprising of selenium, zinc, lycopene, and vitamin C)
  Interventions: Drug: Antioxidant

INTERVENTIONS:
Drug: Paxlovid — This adaptive platform trial will assess therapeutics for SARS-CoV-2 in out-patient settings. The first intervention arm is Paxlovid.
  Arms: Paxlovid
Drug: Antioxidant — Antioxidant therapy (comprising of selenium, zinc, lycopene, and vitamin C)
  Arms: Antioxidant Therapy - Intervention (arm 3)

SUMMARY:
CanTreatCOVID is an open-label, individually randomized, multi-centre, national trial. CanTreatCOVID aims to establish an adaptive platform trial aimed at evaluating the clinical- and cost-effectiveness, practical challenges, and outcomes of therapeutics for SARS-CoV-2 for non-hospitalized patients in Canada. Participants will be randomized to receive usual care (i.e. supportive care and symptom relief) or a study therapeutic, which will be determined by the Canadian COVID-19 Out-Patient Therapeutics Committee. The primary outcomes being evaluated is hospitalization and/or death at 28 days, as well as time to recovery.

DETAILED DESCRIPTION:
While public health measures and vaccines have reduced the impact of SARS-CoV-2 on hospitalization and death, most scientists predict this virus will become endemic and new variants will continue to emerge. Effective and affordable therapeutics for SARS-CoV-2 that can be easily used in community settings are needed to accelerate recovery, prevent hospitalizations and deaths, and to minimize the development of post-acute sequelae of SARS-CoV-2 ("long COVID"). Most randomized controlled trials (RCT) of therapeutics to date have included participants who have not been vaccinated and who did not have previous infections. The Canadian Adaptive Platform Trial of Treatments for COVID in Community Settings (CanTreatCOVID) will evaluate the clinical effectiveness and cost-effectiveness of therapeutics for SARS-CoV-2 in non-hospitalized patients. Adaptive platform trials (APTs) are designed to compare multiple therapies in an efficient manner and allow us to respond to the dynamic nature of the COVID-19 pandemic. Therapeutics to be evaluated will be identified through a transparent Canadian COVID-19 Out-Patient Therapeutics Committee. The co-primary outcomes are all-cause hospitalization and/or death at 28 days as well as time to recovery, and key secondary outcomes include, symptom severity, incidence of post-acute sequelae of SARS-CoV-2, quality of life, and cost-effectiveness of each therapeutic. CanTreatCOVID uses numerous approaches to recruit participants to the study, including a multi-faceted public communication strategy and outreach through primary care, out-patient clinics, and EDs.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years and older or 18-49 with 1 or more chronic high-risk medical conditions, and/or immunosuppression: chronic respiratory disease (including COPD, cystic fibrosis and asthma requiring at least daily use of preventative and/or reliever medication); chronic heart or vascular disease; chronic kidney disease; chronic liver disease; chronic neurological disease (including dementia, stroke, epilepsy); severe and profound learning disability; Down's syndrome; diabetes (Type 1 or Type 2); immunosuppression: primary (e.g. inherited immune disorders resulting from genetic mutations) or secondary due to disease or treatment (e.g. sickle cell, HIV, cancer, chemotherapy); solid organ, bone marrow and stem cell transplant recipients; morbid obesity (BMI >35); severe mental illness; care home resident.
* Confirmed SARS-CoV-2 by nucleic acid testing or rapid antigen testing with proof of a positive test provided via a picture of the result
* Able to be enrolled and begin the study therapeutic within 5 days of onset of symptoms associated with SARS-CoV-2 infection

Exclusion Criteria:

* Admitted to hospital or in an ED for more than 24 hours
* Previously randomized to CanTreatCOVID
* Currently participating in a clinical trial of a therapeutic agent for acute SARS-CoV-2 infection that is not/suspected not compatible with the study therapeutics
* Already taking a study therapeutic or contraindication to a study therapeutic
* Inability for participant or caregiver to provide informed consent

Paxlovid Exclusion Criteria include:

* History of clinically significant hypersensitivity to the active substances in Paxlovid™ (nirmatrelvir /ritonavir) or to any of its excipients.
* Patients with known rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption.
* Patients with known current severe liver impairment (characterized by severe ascites, encephalopathy, jaundice, or prolonged INR. People with liver disease without any of these features are eligible).
* Is a recipient of a solid organ transplant and taking immunosuppressant medications.
* Patients with known moderate or severe renal disease (defined as CKD stage 3, 4 or 5 or current acute kidney injury or most recent eGFR in the past 6 months <60 ml/min).
* Currently taking Paxlovid™.
* Clinical requirement to continue taking a drug which is contraindicated or not recommended for administration with Paxlovid™ in the context of CanTreatCOVID or is taking a drug which in the opinion of the investigator would put the subject at unacceptable risk.
* Has a known or suspected pregnancy.
* Is breastfeeding.
* Is of childbearing potential and is not willing to use a highly effective contraceptive

Antioxidant Exclusion Criteria include:

* Has a known or suspected pregnancy.
* Is breastfeeding.
* Is of childbearing potential and is not willing to use a highly effective contraceptive.
* Has allergy or intolerance to selenium, zinc, lycopene, vitamin C, ascorbyl palmitate, hypromellose, microcrystalline cellulose, or sodium stearyl fumarate
* Is taking warfarin as a preventive measure.
* Has advanced chronic kidney disease (CKD stage 3: eGFR ≥30 to <60 mL/min, and severe renal impairment (eGFR <30 ml/min, CKD stage 4-5)
* Has liver disease awaiting transplantation.
* Has a history of calcium oxalate kidney stones.
* Has a diagnosis of head and neck cancer within the past 5 years
* Has medical history of non-melanoma skin cancer
* Is taking selenium (≥300ug/day), zinc (≥40mg/day), lycopene (≥45mg/day), and vitamin C (≥1500mg/day) supplements at baseline
* Is consuming omega-3 fatty acids at baseline and is unwilling to stop during the intervention period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 797 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-06-28 (Estimated)

PRIMARY OUTCOMES:
All-cause hospitalization or death rate | Day 28

SECONDARY OUTCOMES:
Time to recovery | Days 0-14
  Defined as the first instance that a participant reports feeling fully recovered after enrolment
Symptom severity | Days 0-28
  Symptoms severity will be assessed using the questions: "How well are you feeling today? Please rate how you are feeling now using a scale of 1 - 4, where 1 is no symptoms, and 4 is very severe symptoms" and by rating symptoms, if present, as "No problem, mild problem, moderate problem, or major problem."
Rate of Post-acute sequelae of SARS-CoV-2 | 90 days and 36 weeks
Quality of life measurement (EQ-5D-5L) | Baseline, 21 days, 28 days, 90 days, and 36 weeks
  Measured by EQ-5D-5L questionnaire on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. This scale is numbered from 0 to 100. 100 means the best health you can imagine. 0 means the worst health you can imagine
Early discontinuation and severe adverse events | Days 0-28
Treatment costs | 12 and 24 months
  Cost-utility analysis will be calculated as the incremental cost per QALY gained.

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - The Governors of the University of Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - The University of Manitoba, Winnipeg, Manitoba
  - Eastern Health Newfoundland and Labrador, St. John's, Newfoundland and Labrador
  - Unity Health Toronto, Toronto, Ontario
  - The Research Institute of the McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Our team is dedicated to making data accessible to researchers upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: End of study (TBD) and upon request until 15yrs after study completion.
Access Criteria: Study PI
URL: https://upstreamlab.org

REFERENCES:
- [Derived] Hosseini B, Condon A, da Costa BR, Daley P, Greiver M, Juni P, Lee TC, McBrien K, McDonald EG, Murthy S, Selby P, Andrew M, Aubrey-Bassler K, Barber D, Barrett B, Butler CC, Crampton N, Dahrouge S, Damji A, Fowler R, Garies S, Hudon C, Hulme J, Isenor J, Jenkins DJA, Lall R, LeBlanc A, Leong C, Little P, Lofters A, Logsetty S, Lother S, Lussier MT, Maclaren L, Mangin D, Marshall EG, Marshall JC, McCracken R, Moineddin R, Orava B, Paquette JS, Park JJH, Persaud N, Rac VE, Ramsden VR, Rayner J, Sanchez-Ramirez DC, Saxinger L, Shi H, Singer A, Spiwak R, Srivastava A, Sud A, Tarride JE, Telner D, Upshur REG, Walji S, Walsh R, Wilchesky M, Wong ST, Wood B, Zarychanski R, Zelek B, Keynan Y, Piszczek J, Warshafsky D, Pinto AD. Canadian Adaptive Platform Trial of Treatments for COVID in Community Settings (CanTreatCOVID): protocol for a randomised controlled adaptive platform trial of treatments for acute SARS-CoV-2 infection in community settings. BMJ Open. 2025 Aug 3;15(8):e097134. doi: 10.1136/bmjopen-2024-097134. PMID 40754325
- See also: Related Info — https://cantreatcovid.org/